CLINICAL TRIAL: NCT04542941
Title: Assessment of Safety and Efficacy of COVID-19 Convalescent Plasma for Treatment of COVID-19 in Adults in Uganda; A Randomised Controlled Trial
Brief Title: Assessment of Safety and Efficacy of CCP
Acronym: COVIDIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: Uganda Blood Transfusion Services (Unknown); Joint Clinical Research Center (Other); Uganda Peoples Defence Forces Medical Services (Unknown); Mulago Hospital, Uganda (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCP
Record Dates: First submitted 2020-08-31; First posted 2020-09-09 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Intervention Model Description: This study will be a prospective randomized two arm open label clinical trial. Patients with confirmed COVID-19 who meet the study eligibility criteria will be randomized to receive either CCP in addition to standard of care therapy or standard of care therapy alone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Active Comparator): The participants will receive COVID Convalescent Plasma in addition to the standard of care received by all COVID 19 patients
  Interventions: Biological: COVID Convalescent Plasma
- Control arm (No Intervention): The participants under this arm will receive the COVID 19 standard of care

INTERVENTIONS:
Biological: COVID Convalescent Plasma — Plasma collected from recovered COVID 19 individuals
  Arms: Intervention arm

SUMMARY:
Currently there are no proven treatments or vaccines for COVID-19 and care of the COVID patients is largely supportive involving treatment of symptoms such as fever with antipyretics, secondary bacterial chest infection with antibiotics and meticulous management of comorbid conditions.

Several repurposed and new drugs have been investigated for treatment of COVID-19, however, none have been confirmed to be efficacious. These drugs include the antimalarials (chloroquine and hydroxychloroquine), antivirals such as remdesivir and favipiravir and antiretroviral combination therapies such lopinavir/ritonavir.

There is emerging evidence to support the use of COVID convalescent plasma for the treatment of COVID-19. There is need to leverage the blood transfusion services in countries and this is beginning to happen on the continent.

DETAILED DESCRIPTION:
Currently there are no proven treatments for COVID-19 and current standard therapy is supportive care with oxygen supplementation and treatment of symptoms. While treatments are being investigated in the Western world, it is likely that these data will take several months to become available and if proven to be efficacious, access in most of the low-income countries will be limited due to the high global demand and exorbitant costs.

In this study, the investigators aim to assess the safety and efficacy of use of CCP for treatment of adults with COVID-19 in Uganda.

The investigators hypothesise that administration of CCP to patients with positive SARS-CoV-2 RT PCR leads to earlier time to viral clearance compared to the standard of care.

Objectives:

General objective The overall objective of this project is to assess the safety and efficacy of COVID-19 convalescent plasma in the treatment of COVID-19 in Uganda.

Primary objective

1. To determine the efficacy of COVID-19 Convalescent Plasma, as measured by time to RT-PCR negativity of COVID-19 patients treated with COVID-19 Convalescent Plasma.

Secondary objectives

1. To assess the safety of COVID-19 Convalescent Plasma in the treatment of COVID-19 patients in Uganda
2. To document the time to symptom decrease of patients with positive SARS-CoV-2 RT PCR treated with CCP compared to those on standard of care
3. To assess the ability of CCP therapy to stop progression to severe/critical forms of disease This study will be a prospective randomized two arm open label clinical trial. Patients with confirmed COVID-19 who meet the study eligibility criteria will be randomized to receive either CCP in addition to standard of care therapy or standard of care therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Adults with documented laboratory RT PCR confirmed SAR-CoV-2 infection
* Patients able to provide informed consent. In the event that the patient cannot provide consent e.g. they are severely sick, the next of kin or legal surrogate decision make

Exclusion Criteria:

* Prior diagnosis of IgA deficiency
* Inability to return for post discharge follow up

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Time to viral clearance (RT-PCR negativity) | 28 days
  The primary end point will be time to viral clearance (RT-PCR negativity).

SECONDARY OUTCOMES:
Time to symptom resolution | 28 days
  time to symptom resolution (resolution of the major COVID-19 symptoms of fever, cough, and shortness of breath, rhinorrhea and fatigue)
Time to severe/critical disease | 28 days
  Time to clinical improvement as evidenced by the modified ordinal scale for clinical improvement which has 8 states (not hospitalised and not on Oxygen therapy, hospitalised and on oxygen therapy, hospitalised no oxygen therapy, oxygen therapy by nasal prongs (<5l/min), oxygen therapy by mask, SFM or NRM (>10l/min), intubation and mechanical ventilation, ventilation plus additional organ support, death
Number of participants reporting an adverse event as evidenced by clinical manifestations | 28 days
  Safety of convalescent plasma as determined by clinical manifestations eg Skin or mucous membrane manifestations, respiratory compromise, Decrease in systolic blood pressure to <90 mmHg or >30% decrease from baseline or a diastolic drop of >30% from baseline, Tachycardia with an increase in resting heart rate to >130 bpm; or bradycardia <40 bpm that is associated with dizziness, nausea or feeling faint, Any other symptom which the good clinical judgment of the physician warrants halting the infusion (i.e., rapid onset of gastrointestinal symptoms, etc.)

CONTACTS AND LOCATIONS:
Locations (1):
- Mulago Specialised Hospital, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No
Arrangments to enable sharing of de-identified data will be instituted by the research team.

REFERENCES:
- [Derived] Kirenga B, Byakika-Kibwika P, Muttamba W, Kayongo A, Loryndah NO, Mugenyi L, Kiwanuka N, Lusiba J, Atukunda A, Mugume R, Ssali F, Ddungu H, Katagira W, Sekibira R, Kityo C, Kyeyune D, Acana S, Aanyu-Tukamuhebwa H, Kabweru W, Nakwagala F, Bagaya BS, Kimuli I, Nantanda R, Buregyeya E, Byarugaba B, Olaro C, Mwebesa H, Joloba ML, Siddharthan T, Bazeyo W. Efficacy of convalescent plasma for treatment of COVID-19 in Uganda. BMJ Open Respir Res. 2021 Aug;8(1):e001017. doi: 10.1136/bmjresp-2021-001017. PMID 34376401